CLINICAL TRIAL: NCT05652881
Title: Does Joint Lavage Reduce Intraarticular Inflammation in High-energy Tibial Pilon Fractures?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Benjamin Wheatley, Assistant Clinical Professor, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-14283; R21AR081008 (NIH)
Record Dates: First submitted 2022-11-28; First posted 2022-12-15 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Post-traumatic; Arthrosis; Tibial Fractures; Post-Traumatic Osteoarthritis of Ankle
MeSH Terms: conditions — Osteoarthritis; Tibial Fractures

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Cytokine analysis and radiographic assessment will be performed by a blinded assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Standard of care treatment for axially unstable tibial pilon fracture will include temporary external fixation followed by delayed definitive fixation. Arthrocentesis of the injured and uninjured ankles will be performed at the time of initial temporary external fixation and again at the time of definitive fixation.
- Intervention (Experimental): Additional intra-articular joint lavage with 1L normal saline will be performed at the time of initial temporary external fixation in addition to standard of care treatment.
  Interventions: Procedure: Joint Lavage

INTERVENTIONS:
Procedure: Joint Lavage — An arthrotomy will be made at the time of temporary external fixation and 1L normal saline will be used to irrigate the ankle joint.
  Arms: Intervention

SUMMARY:
High-energy tibial pilon fractures have historically been associated with poor outcomes largely due to the elevated risk of severe post-traumatic arthritis. Intraarticular fractures result in a pro-inflammatory hemarthrosis that may further exacerbate the chondral damage that was sustained due to the original injury. This project will study the effect of joint lavage on the concentration of inflammatory cytokines in the ankle following a high-energy tibial pilon fracture and the resultant effect on short-term patient outcomes.

DETAILED DESCRIPTION:
High-energy pilon fractures are associated with an increased risk of post-traumatic arthritis and poor patient outcomes. The risk of arthritis is over 25% in many series and can be upwards of 50% in more highly comminuted fracture patterns. Intraarticular fractures result in an increase in the synovial concentrations of inflammatory cytokines and matrix metalloproteinases. Animal models have demonstrated the irreversible damage a persistent hemarthrosis may have on cartilage viability suggesting that prolonged exposure to blood in this highly pro-inflammatory milieu may further exacerbate the chondral damage from the initial injury. However, the impact of these local inflammatory processes on the risk of post-traumatic arthritis and patient outcomes remain unclear.

The long-term goal of our research is to develop treatment modalities including surgical and pharmaceutical interventions to reduce the risk post-traumatic arthritis and dysfunction following intraarticular fractures. The objective of this study is to determine the effect of ankle joint lavage on the risk of post-traumatic arthritis and patient outcomes following high-energy pilon fractures. First, we will obtain synovial fluid samples from the ankle joint of patients undergoing temporary external fixation of a pilon fracture for cytokine analysis. Then, we will randomize patients to undergo standard treatment with or without ankle joint lavage at the time of external fixation. Patients will undergo repeat synovial fluid analysis at the time of definitive fixation to determine the effect of lavage on the concentration of pro-inflammatory cytokines. Last, patients will be followed for a period of six months after surgery to determine the impact on functional outcomes.

The information generated in this study will substantially add to our understanding of the pathogenesis of post-traumatic arthritis in high-energy pilon fractures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 years or older
* Present with an axially unstable tibial pilon fracture requiring temporary external fixation followed by delayed definitive internal fixation
* Able to give informed consent

Exclusion Criteria:

* Open fractures
* Delayed presentation greater than 72 hours post-injury
* Associated talar body fracture
* Presentation after initial ex-fix placement
* Unreconstructable or unsalvageable joint
* Preexisting ankle arthritis
* Previous ankle surgery
* Contralateral ankle injury
* Age less than 18 years
* Pregnant women
* Individuals who are incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The effect of intraarticular lavage on the synovial concentration of inflammatory cytokines | 2 years
  The concentration of multiple pro-inflammatory cytokines will be measured in both the injured and non-injured extremity at the time of initial temporary external fixation and definitive fixation.

SECONDARY OUTCOMES:
Effect of intraarticular lavage on functional outcomes following high-energy pilon fractures | 6 months
  American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot scores will be collected at 3 and 6 months post-operatively. The AOFAS Ankle-hindfoot score is on a scale of 0-100 with higher scores indicating better function.
Effect of intraarticular lavage on radiographic outcomes following high-energy pilon fractures | 6 months
  We will evaluate radiographs obtained during the first 6 months to determine the presence and severity of post-traumatic arthritis.
Effect of intraarticular lavage on range of motion following high-energy pilon fractures | 6 months
  Range of motion measurements will be obtained at 3 and 6 months post-operatively

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen SH, Wu PH, Lee YS. Long-term results of pilon fractures. Arch Orthop Trauma Surg. 2007 Jan;127(1):55-60. doi: 10.1007/s00402-006-0225-3. Epub 2006 Sep 27. PMID 17004076
- [Background] Pollak AN, McCarthy ML, Bess RS, Agel J, Swiontkowski MF. Outcomes after treatment of high-energy tibial plafond fractures. J Bone Joint Surg Am. 2003 Oct;85(10):1893-900. doi: 10.2106/00004623-200310000-00005. PMID 14563795
- [Background] Sands A, Grujic L, Byck DC, Agel J, Benirschke S, Swiontkowski MF. Clinical and functional outcomes of internal fixation of displaced pilon fractures. Clin Orthop Relat Res. 1998 Feb;(347):131-7. PMID 9520883
- [Background] De-Las-Heras-Romero J, Lledo-Alvarez AM, Lizaur-Utrilla A, Lopez-Prats FA. Quality of life and prognostic factors after intra-articular tibial pilon fracture. Injury. 2017 Jun;48(6):1258-1263. doi: 10.1016/j.injury.2017.03.023. Epub 2017 Mar 22. PMID 28365069
- [Background] Anderson DD, Marsh JL, Brown TD. The pathomechanical etiology of post-traumatic osteoarthritis following intraarticular fractures. Iowa Orthop J. 2011;31:1-20. PMID 22096414
- [Background] Adams SB, Setton LA, Bell RD, Easley ME, Huebner JL, Stabler T, Kraus VB, Leimer EM, Olson SA, Nettles DL. Inflammatory Cytokines and Matrix Metalloproteinases in the Synovial Fluid After Intra-articular Ankle Fracture. Foot Ankle Int. 2015 Nov;36(11):1264-71. doi: 10.1177/1071100715611176. Epub 2015 Oct 8. PMID 26449389
- [Background] Adams SB, Reilly RM, Huebner JL, Kraus VB, Nettles DL. Time-Dependent Effects on Synovial Fluid Composition During the Acute Phase of Human Intra-articular Ankle Fracture. Foot Ankle Int. 2017 Oct;38(10):1055-1063. doi: 10.1177/1071100717728234. Epub 2017 Sep 11. PMID 28891711
- [Background] Adams SB, Leimer EM, Setton LA, Bell RD, Easley ME, Huebner JL, Stabler TV, Kraus VB, Olson SA, Nettles DL. Inflammatory Microenvironment Persists After Bone Healing in Intra-articular Ankle Fractures. Foot Ankle Int. 2017 May;38(5):479-484. doi: 10.1177/1071100717690427. Epub 2017 Jan 31. PMID 28142266
- [Background] Wahl EP, Lampley AJ, Chen A, Adams SB, Nettles DL, Richard MJ. Inflammatory cytokines and matrix metalloproteinases in the synovial fluid after intra-articular elbow fracture. J Shoulder Elbow Surg. 2020 Apr;29(4):736-742. doi: 10.1016/j.jse.2019.09.024. Epub 2019 Nov 26. PMID 31784384
- [Background] Pham TM, Frich LH, Lambertsen KL, Overgaard S, Schmal H. Elevation of Inflammatory Cytokines and Proteins after Intra-Articular Ankle Fracture: A Cross-Sectional Study of 47 Ankle Fracture Patients. Mediators Inflamm. 2021 Jan 8;2021:8897440. doi: 10.1155/2021/8897440. eCollection 2021. PMID 33505222
- [Background] van Meegeren ME, Roosendaal G, Jansen NW, Lafeber FP, Mastbergen SC. Blood-Induced Joint Damage: The Devastating Effects of Acute Joint Bleeds versus Micro-Bleeds. Cartilage. 2013 Oct;4(4):313-20. doi: 10.1177/1947603513497569. PMID 26069675
- [Background] Ni GX, Zhou YZ, Chen W, Xu L, Li Z, Liu SY, Lei L, Zhan LQ. Different responses of articular cartilage to strenuous running and joint immobilization. Connect Tissue Res. 2016;57(2):143-51. doi: 10.3109/03008207.2015.1117457. Epub 2015 Dec 2. PMID 26631363
- [Background] Campbell TM, Reilly K, Laneuville O, Uhthoff H, Trudel G. Bone replaces articular cartilage in the rat knee joint after prolonged immobilization. Bone. 2018 Jan;106:42-51. doi: 10.1016/j.bone.2017.09.018. Epub 2017 Sep 30. PMID 28974461
- [Background] Nomura M, Sakitani N, Iwasawa H, Kohara Y, Takano S, Wakimoto Y, Kuroki H, Moriyama H. Thinning of articular cartilage after joint unloading or immobilization. An experimental investigation of the pathogenesis in mice. Osteoarthritis Cartilage. 2017 May;25(5):727-736. doi: 10.1016/j.joca.2016.11.013. Epub 2016 Dec 1. PMID 27916560
- [Background] Al-Ashhab ME. Primary Ankle Arthrodesis for Severely Comminuted Tibial Pilon Fractures. Orthopedics. 2017 Mar 1;40(2):e378-e381. doi: 10.3928/01477447-20161202-04. Epub 2016 Dec 15. PMID 27942740
- [Background] Ho B, Ketz J. Primary Arthrodesis for Tibial Pilon Fractures. Foot Ankle Clin. 2017 Mar;22(1):147-161. doi: 10.1016/j.fcl.2016.09.010. Epub 2016 Dec 20. PMID 28167059
- [Background] Thomas NP, Wu WJ, Fleming BC, Wei F, Chen Q, Wei L. Synovial inflammation plays a greater role in post-traumatic osteoarthritis compared to idiopathic osteoarthritis in the Hartley guinea pig knee. BMC Musculoskelet Disord. 2017 Dec 29;18(1):556. doi: 10.1186/s12891-017-1913-6. PMID 29284451
- [Background] Catterall JB, Stabler TV, Flannery CR, Kraus VB. Changes in serum and synovial fluid biomarkers after acute injury (NCT00332254). Arthritis Res Ther. 2010;12(6):R229. doi: 10.1186/ar3216. Epub 2010 Dec 31. PMID 21194441
- [Background] Wei L, Fleming BC, Sun X, Teeple E, Wu W, Jay GD, Elsaid KA, Luo J, Machan JT, Chen Q. Comparison of differential biomarkers of osteoarthritis with and without posttraumatic injury in the Hartley guinea pig model. J Orthop Res. 2010 Jul;28(7):900-6. doi: 10.1002/jor.21093. PMID 20108346
- [Background] Boutet MA, Najm A, Bart G, Brion R, Touchais S, Trichet V, Layrolle P, Gabay C, Palmer G, Blanchard F, Le Goff B. IL-38 overexpression induces anti-inflammatory effects in mice arthritis models and in human macrophages in vitro. Ann Rheum Dis. 2017 Jul;76(7):1304-1312. doi: 10.1136/annrheumdis-2016-210630. Epub 2017 Mar 13. PMID 28288964
- [Background] Zhang Y, Qian X, Yang X, Niu R, Song S, Zhu F, Zhu C, Peng X, Chen F. ASIC1a induces synovial inflammation via the Ca2+/NFATc3/ RANTES pathway. Theranostics. 2020 Jan 1;10(1):247-264. doi: 10.7150/thno.37200. eCollection 2020. PMID 31903118
- [Background] Holzer N, Salvo D, Marijnissen AC, Vincken KL, Ahmad AC, Serra E, Hoffmeyer P, Stern R, Lubbeke A, Assal M. Radiographic evaluation of posttraumatic osteoarthritis of the ankle: the Kellgren-Lawrence scale is reliable and correlates with clinical symptoms. Osteoarthritis Cartilage. 2015 Mar;23(3):363-9. doi: 10.1016/j.joca.2014.11.010. Epub 2014 Nov 15. PMID 25463444
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Madeley NJ, Wing KJ, Topliss C, Penner MJ, Glazebrook MA, Younger AS. Responsiveness and validity of the SF-36, Ankle Osteoarthritis Scale, AOFAS Ankle Hindfoot Score, and Foot Function Index in end stage ankle arthritis. Foot Ankle Int. 2012 Jan;33(1):57-63. doi: 10.3113/FAI.2012.0057. PMID 22381237
- [Background] Lau JT, Mahomed NM, Schon LC. Results of an Internet survey determining the most frequently used ankle scores by AOFAS members. Foot Ankle Int. 2005 Jun;26(6):479-82. doi: 10.1177/107110070502600609. PMID 15960915